CLINICAL TRIAL: NCT03415087
Title: Sequential Intrathecal Injection of Fentanyl and Hyperbaric Bupivacaine at Different Rates; Does it Make Difference?
Brief Title: Sequential Intrathecal Injection of Fentanyl and Hyperbaric Bupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: R47
Record Dates: First submitted 2017-12-24; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Elective Caesarean Section
MeSH Terms: interventions — Fentanyl; Analgesics, Opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sequential intrathecal injection of fentanyl and bupivacaine (Active Comparator): intrathecal injection drug: fentanyl 25 μg (0.5 ml), IV,once drug: hyperbaric bupivacaine 0.5%10 mg IV,once both syringes were injected slowly sequentially
  Interventions: Procedure: sequential intrathecal injection; Drug: hyperbaric bupivacaine; Drug: fentanyl
- rapid sequential intrathecal injection of fentanyl and bupiva (Experimental): intrathecal injection drug: fentanyl 25 μg (0.5 ml), IV, injected rapidly and mixed by CSF, once drug: hyperbaric bupivacaine 0.5%10 mg IV injected slowly once.
  Interventions: Procedure: sequential intrathecal injection; Drug: hyperbaric bupivacaine; Drug: fentanyl

INTERVENTIONS:
Procedure: sequential intrathecal injection — intrathecal injection of fentanyl and hyperbaric bupivacaine
  Other Names: sequential spinal anaesthesia
Drug: hyperbaric bupivacaine — intrathecal injection of intrathecal bupivacaine
  Other Names: heavy marcaine
Drug: fentanyl — intrathecal injection of fentanyl
  Other Names: opioid

SUMMARY:
56 Parturients, aged 18-40 year, undergoing elective CS were randomly assigned to receive sequential intrathecal injection of fentanyl and hyperbaric bupivacaine at the same rate (normal sequential) NS or a rapid intrathecal injection of fentanyl followed by slow injection of hyperbaric bupivacaine (rapid sequential) RS. Time of first rescue analgesia, Dose of rescue analgesics, degree of postoperative pain, incidence of hypotension, hypotension duration, ephedrine dose, spinal anaesthesia related complications and failed block were recorded.

DETAILED DESCRIPTION:
56 ASA physical status I, II Parturients, aged 18-40 year, undergoing elective CS were randomly assigned to receive sequential intrathecal injection of fentanyl and hyperbaric bupivacaine at the same rate through a 5ml syringe each (NS (normal sequential), n 28) or a rapid intrathecal injection of fentanyl through an insuline syringe followed by slow injection of hyperbaric bupivacaine through a 5ml syringe RS (rapid sequential), n 28). Onset of sensory block (T6 level), highest level of sensory block, time of first rescue analgesia, Dose of rescue analgesics, degree of postoperative pain by VAS 6H postoperative, Onset of motor block (Bromage scale0>3), duration of motor block (return to Bromage 0), incidence of hypotension, hypotension duration, ephedrine dose, spinal anaesthesia related complications as nausea, vomiting, pruritis, shivering and failed block were recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II
* Parturients aged from 18-40 years old
* scheduled for elective CS

Exclusion Criteria:

* parturients with complicated pregnancy as (preeclampsia, pregnancy induced HTN, gestational Diabetes, abnormal placenta (placenta previa), multiple gestation),
* BMI greater than 35 or less than 22,
* major systemic disease (cardiac, renal, liver),
* need for emergency CS,
* having allergy to drugs used in the study,
* having contraindication for spinal anaesthesia or
* refused regional anaesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — females undergoing CS
Enrollment: 56 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | 2-5 hours
  technique provides prolonged post operative analgesia

SECONDARY OUTCOMES:
incidence of hypotension | 30 minutes
  note if hypotension occurs